CLINICAL TRIAL: NCT01221064
Title: Prospective Randomised Clinical Trial Comparing the Effect of Early and Late Drainage Removal in Female Patients After Radical Mastectomy With Axillary Clearance
Brief Title: Effect of Early vs Late Drainage Removal in Women After Radical Mastectomy With Axillary Clearance
Acronym: CHLONKA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Jacek Zielinski, Assistant Profesor, Medical University of Gdansk
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MUGSO-001
Record Dates: First submitted 2010-10-06; First posted 2010-10-14 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Axillary clearance; lymphorrhoea
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early drainage removal (Other): Patients randomised to early drainage removal arm will have the drain removed in postoperative day 1. Lymph will be punctured on a regular basis
  Interventions: Procedure: Early drainage removal
- Late drainage removal (Other): Patients randomised to late drainage removal arm will have the drains kept until total daily drainage is 30ml and then removed
  Interventions: Procedure: Late drainage removal

INTERVENTIONS:
Procedure: Early drainage removal — Drainage will be removed in postoperative day 1
  Arms: Early drainage removal
Procedure: Late drainage removal — Drains will be kept until daily drainage is 30ml and then removed
  Arms: Late drainage removal

SUMMARY:
The aim of the study is to assess whether early drainage removal in patients with less than 150ml of lymph in postoperative day 1 can reduce total lymphorrhoea

DETAILED DESCRIPTION:
Patients with early drainage removal will be compared with patients in whom drainage will be kept until daily lymphorrhoea is 30ml

ELIGIBILITY:
Inclusion Criteria:

* Stage IIA and IIB breast cancer treated with radical mastectomy
* Obtaining informed consent
* Total amount of lymph in postoperative day 1 <150ml

Exclusion Criteria:

* Stage I, III-IV breast cancer
* History of benign breast neoplasm or malignant disease of any origin
* Any breast surgery in the past
* Weight <50kg

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Total lymph volume and time | 3 months
  Assessment of total lymph volume and lymphorrhoea time up to 3 months after the surgery

SECONDARY OUTCOMES:
Post operative pain assessment | 30 days
  Post operative pain assessment using VAS (Visual Analogue Scale) scale until 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Janusz Jaśkiewicz, MD, PhD, Study Director — Medical University of Gdansk; Jacek Zielinski, MD, PhD, Principal Investigator — Medical University of Gdansk
Locations (1):
- Medical University of Gdansk, Department of Surgical Oncology, Gdansk, Pomeranian Voivodeship, Poland